CLINICAL TRIAL: NCT01915875
Title: Impact of Global Care of the Pain at Chronic Painful Patients Affected by Cystic Fibrosis
Acronym: MUCO-SOPHRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Fondation de France (Other); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: P070706; 2008-A01575-50 (Other: EudraCT Number)
Record Dates: First submitted 2012-07-20; First posted 2013-08-05 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis-pain-sophrology
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- sophrology sessions (Experimental): The sophrology is a dynamic method of physical and psychical relaxation
  Interventions: Other: sophrology sessions at home

INTERVENTIONS:
Other: sophrology sessions at home — The sophrology is a dynamic method of physical and psychical relaxation

SUMMARY:
The purpose of this study is to evaluate the impact of the global approach to the pain in cystic fibrosis patients with chronic or intermittent pain. The patients will receive in addition to an usual pharmacological and psychological management, sophrology sessions at home. The results of this study will provide a new strategy of management of the patient's pain.

DETAILED DESCRIPTION:
The majority of cystic fibrosis patients have chronic or intermittent pains. These pains have important consequences on the quality of life. Currently, the treatment is essentially pharmacological (essentially paracetamol) but it is not enough in presence of of visual analogue scale (VAS) >4. In the study, the patients will receive in addition to an usual pharmacological and psychological management, sophrology sessions at home. The sophrology is a dynamic method of physical and psychical relaxation. This aims are to decrease the pain, to decrease the anxiety and to improve the everyday life. This study will provide a new global strategy of the management of the patients' pain.

ELIGIBILITY:
Inclusion Criteria:

* Cystic fibrosis patients defined by a test sweat and / or 2 pathogenic mutations
* Patients over 10 years
* Patients with pain symptoms (VAS> 4) recurrent (> 4 episodes / month) or permanent since more than 6 months
* Agreement of patients, and parents (for children) for sophrology sessions conducted at home.
* Patient affiliated to social security

Exclusion Criteria:

* Transplant patients or placed on a waiting list transplantation
* Patients had a patient-support by techniques hypnosis or relaxation therapy, during or within 3 months.
* Patients enrolled in another research interventional protocol.
* Women without contraception or pregnant.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-02-15 (Actual); Primary Completion 2014-11-19 (Actual); Study Completion 2014-11-19 (Actual)

PRIMARY OUTCOMES:
Change of maximum VAS | 6 months
  Change of maximum VAS for the site presenting a max VAS in the month following the inclusion.

SECONDARY OUTCOMES:
number of paroxystic episodes | 6 months
  Change of the number of paroxystic episodes
intensity of maximum VAS of the painful episodes | 6 months
  Change of the intensity of maximum VAS of the painful episodes between the month following the inclusion and last month of the study (for all the sites)
Improvement of the quality of life | 6 months
  Questionnaire of Quality of life CFQ 14 + and CHILD: physical functioning, vitality, body image and respiratory symptoms
BMI | 6 months
  improvement of the BMI,
VEMS | 6 months
  improvement of the VEMS
CVF | 6 months
  improvement of the CVF
SaO2 | 6 months
  improvement of the SaO2

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Sermet, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- hôpital Necker Enfants malades, Paris, France